CLINICAL TRIAL: NCT06321952
Title: A Comparison of Accuracy and Functional Outcome Between Robotic Assisted Surgery and Gyroscopic Based Instrument in Primary Total Knee Arthroplasty
Brief Title: Comparison of Accuracy and Functional Outcome Between Robotic and Gyroscopic Assisted Surgery in Primary TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTanareesuchoti
Record Dates: First submitted 2024-02-12; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Knee Arthropathy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROSA robotic assist TKA (Active Comparator): ROSA robotic assist TKA
  Interventions: Device: ROSA robotic assist TKA
- iassist TKA (Active Comparator): iassist TKA
  Interventions: Procedure: iassist TKA

INTERVENTIONS:
Device: ROSA robotic assist TKA — total knee replacement with ROSA robotic assist
  Other Names: iassist TKA
  Arms: ROSA robotic assist TKA
Procedure: iassist TKA — total knee replacement with iassist
  Arms: iassist TKA

SUMMARY:
A randomized controlled trial was conducted with 72 participants who had moderate knee osteoarthritis (Kellgren and Lawrence grade 2-3). The patients were randomly assigned to either the robotic-assisted or gyroscopic-assisted group. Baseline characteristics, including age, body mass index, length of stay, and estimated blood loss, were recorded. The primary outcome measure was the accuracy of the hip knee angle, measured by scannogram film preoperatively and postoperatively at 3 months. Secondary outcomes included functional outcomes (KOOS, Oxford knee score, EQ-5D-5L, range of motion) assessed preoperatively and postoperatively at 3 months, as well as at 6 months postoperatively.

DETAILED DESCRIPTION:
Introduction: Primary total knee arthroplasty is considered the gold standard treatment for end-stage osteoarthritis of the knee. The primary objective of this surgical procedure is to restore mechanical alignment. At Siriraj Hospital, we employ technology to enhance the accuracy of our surgical procedures. The purpose of this study is to compare the accuracy of robotic-assisted surgery (ROSA) and gyroscope-based surgery in primary total knee arthroplasty.

Methods: A randomized controlled trial was conducted with 72 participants who had moderate knee osteoarthritis (Kellgren and Lawrence grade 2-3). The patients were randomly assigned to either the robotic-assisted or gyroscopic-assisted group. Baseline characteristics, including age, body mass index, length of stay, and estimated blood loss, were recorded. The primary outcome measure was the accuracy of the hip knee angle, measured by scannogram film preoperatively and postoperatively at 3 months. Secondary outcomes included functional outcomes (KOOS, Oxford knee score, EQ-5D-5L, range of motion) assessed preoperatively and postoperatively at 3 months, as well as at 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* primary osteoarthritis knee with indicated for total knee replacement
* age equal or more than 55 years old

Exclusion Criteria:

* revision surgery
* deformity greater than 15º
* Intra/Post operative complication

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
accuracy of Robotic Assisted Surgery and Gyroscopic Based Instrument | preoperative and postoperative 3months
  accuracy of the hip knee angle, measured by scannogram film preoperatively and postoperatively at 3 months

SECONDARY OUTCOMES:
Functional Outcome of Robotic Assisted Surgery and Gyroscopic Based Instrument | preoperative and postoperative 3months and 6months
  functional outcomes (KOOS score) score 0-100 in each domain of 4 domains 0=worst, 100=good
Functional Outcome of Robotic Assisted Surgery and Gyroscopic Based Instrument | preoperative and postoperative 3months and 6months
  functional outcomes (Oxford knee score) score 0-48 0=worst, 48=good
Functional Outcome of Robotic Assisted Surgery and Gyroscopic Based Instrument | preoperative and postoperative 3months and 6months
  functional outcomes (EQ-5D-5L) score 5-25, score5=good, 25=worst
Functional Outcome of Robotic Assisted Surgery and Gyroscopic Based Instrument | preoperative and postoperative 3months and 6months
  functional outcomes (range of motion)

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided